CLINICAL TRIAL: NCT03257618
Title: Quality of Life and Neurocognitive Functioning in Diffuse Low-grade Glioma (TEMOIN)
Brief Title: Quality of Life and Neurocognitive Functioning
Acronym: TEMOIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICM-URC2016-32
Record Dates: First submitted 2017-08-16; First posted 2017-08-22 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Temozolomide; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temozolomide (Experimental): Treatment with TMZ will be given orally according to standard practices. The therapeutic schedule will be left at the investigator's discretion.
  Patients will be followed every 3 months during the treatment period, at the end of the treatment with TMZ, 6 months after the end of TMZ, and then annually until tumor progression.
  Interventions: Drug: Temozolomide; Other: QoL, neurocognitive and psycholpathological assessment

INTERVENTIONS:
Drug: Temozolomide — Treatment with TMZ will be given orally according to standard practices. The therapeutic schedule will be left at the investigator's discretion.
  Patients will be followed every 3 months during the treatment period, at the end of the treatment with TMZ, 6 months after the end of TMZ, and then annually until tumor progression.
Other: QoL, neurocognitive and psycholpathological assessment — This assessment will be performed at baseline, at 6 months, 12 months, 18 months, at the end of the treatment with TMZ, 6 months after the end of TMZ

SUMMARY:
Studying QoL in patients DLGG receiving TMZ is complex because of the multiples interactions between tumor characteristics, neurocognitive functioning, treatments, environment and psychopathological context in which these patients experience symptoms. It is, however, important to accurately evaluate these aspects in consideration of the young age, generally preserved QoL at the time of diagnosis, possible implications of the disease on the professional (DLGG patients are often still active), social and familial domain, and relatively long survival of these patients. In the absence of a curative treatment for DLGG, preserving patients' QoL is indeed a major goal.

DETAILED DESCRIPTION:
Diffuse low-grade gliomas (DLGG) (or WHO grade II gliomas, Louis et al., 2007) are rare tumors, with an incidence estimated at 1/105 person-year (Ostrom et al., 2015). They affect young people in their thirties or forties (Capelle et al., 2013). DLGG are characterized by a continuous growth and an unavoidable anaplastic transformation (Mandonnet et al., 2003). Epilepsy is the main presenting mode while neurological deficits are rare at diagnosis due to the brain plasticity allowed by the usually slow growth speed of these tumors. However, frequent alterations in cognitive functions (including mostly memory, executive functioning, and attention) have been described (Racine et al., 2015). The prognosis of DLGG is variable (Pignatti et al., 2002) and overall survival (OS) ranges from 5 years to 15 years according to several factors, including the tumor phenotype, the isocitrate dehydrogenase (IDH) mutation and the 1p19q codeletion, the tumor volume at diagnosis, and the tumor spontaneous growth speed (Capelle et al., 2013).

The prognostic impact of the extent of surgery has now been well demonstrated (Jakola et al., 2012; Duffau 2016) and surgery is now the first treatment option (Soffietti et al., 2010). In unresectable DLGG or in patients with a progressive disease after surgery (with no possibility of a second surgery), several treatment options have been investigated, including radiation therapy (RT) and chemotherapy, but to date the timing and choice of treatment remains controversial. RT can be efficient in DLGG, however, the EORTC 22845 phase III trial found that early RT has no impact on OS compared to late RT, despite an increased progression-free survival (PFS) (van Den Bent et al., 2005). Moreover, some evidence of late decreased neurocognitive functioning has been consistently reported following RT (Klein et al., 2002; Douw et al., 2009). Because of this potential neurotoxicity and the absence of a benefit on OS of early RT, many neuro-oncological teams now only offer RT to patients with a progressive disease after chemotherapy.

Temozolomide (TMZ), an orally administered drug, was shown to be efficient in DLGG, with a good tolerance (Hoang-Xuan et al., 2004; Ricard et al., 2007). However, data regarding the impact of TMZ on neuro-cognitive functioning and quality of life (QoL) are scarce. Only few studies have performed an extensive, longitudinal assessment of cognition and QoL in DLGG patients receiving TMZ (Liu et al., 2009; Blonski et al., 2012; Klein, 2015). Moreover, many studies did not take into account the other factors that can alter the cognition such as the tumor itself, the surgery, seizures, anti-epileptic drugs, but also the premorbid level of cognition and the psychopathological affects such as depression, anxiety, or anger (Klein, 2015). To date, there is only few data on these psychopathological aspects in DLGG patients, either at diagnosis or following chemotherapy or RT.

Studying QoL in patients DLGG receiving TMZ is complex because of the multiples interactions between tumor characteristics, neurocognitive functioning, treatments, environment and psychopathological context in which these patients experience symptoms. It is, however, important to accurately evaluate these aspects in consideration of the young age, generally preserved QoL at the time of diagnosis, possible implications of the disease on the professional (DLGG patients are often still active), social and familial domain, and relatively long survival of these patients. In the absence of a curative treatment for DLGG, preserving patients' QoL is indeed a major goal.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged ≥ 18, no age limit;
* Histologically-proven DLGG;
* Patient receiving TMZ as a first line treatment after surgery, whatever the delay between the surgery and the introduction of TMZ;
* No previous oncologic treatment (except for surgery) for the DLGG;
* Performance status (PS) score ≤ 2;
* Absolute neutrophil count (ANC) ≥ 1500 cells/µL and platelet count ≥ 100 000 cells/µL;
* Total serum bilirubin concentration ≤ 1.5 x the upper limit of normal (ULN);
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase ≤ 2.5 x the ULN;
* Serum creatine concentration ≤ 1.5 x the ULN;
* Negative pregnancy test in women of childbearing potential;
* A signed informed consent obtained before any study specific procedures;
* Patient fluent in French ;
* Patient affiliated to a French social security system

Exclusion Criteria:

* Anaplastic glioma (WHO grade III glioma);
* Impaired neurocognitive functioning defined by a score < 22 at the MoCA evaluation;
* Visual or auditory deficit ;
* Previous chemotherapy for the DLGG;
* Previous RT for the DLGG;
* Known hypersensitivity to any of the study drugs, or excipients in the formulation;
* Hypersensitivity to dacarbazine (DTIC);
* Severe myelosuppression;
* Problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption;
* Legal incapacity or physical, psychological social or geographical status interfering with the patient's ability to sign the informed consent or to terminate the study;
* Pregnant or breastfeeding women;
* Men or women of childbearing potential who are unwilling to employ adequate contraception, from the beginning of the study until 6 months after administration of the last treatment dose;
* Participation in another clinical trial with 30 prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
proportion of patients that consent to participate in the study | through study completion, an average of 5 year
  The participation rate: the proportion of patients that consent to participate in the study among the screened patients.
proportion of included patients that will complete the evaluations at baseline, 6 months and 12 months | through study completion, an average of 5 year
  proportion of included patients that will complete the evaluations at baseline, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: jean pierre bleuse, Study Director — Institut régional du Cancer de Montpellier
Locations (1):
- Institut regional du Cancer - Val d Aurelle, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided